CLINICAL TRIAL: NCT03007277
Title: Evaluation de l'Intervention Des Services de Protection Maternelle et Infantile de 11 départements français Ayant bénéficié d'un référentiel Commun d'Intervention à Domicile (Projet Panjo : Promotion de la Santé et de l'Attachement Des Nouveau-nés et de Leurs Jeunes Parents : un Outil de Renforcement Des Services de PMI)
Brief Title: Evaluation of the French Maternal and Child Protection Services From 11 French Territories That Have Received Common Intervention Guidelines
Acronym: PANJO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Agence des Nouvelles Interventions Sociales et de Santé (Other)
Collaborators: Institut national de prevention et d'education pour la sante (Other Government); Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Thomas Saias, Professeur, L'Agence des Nouvelles Interventions Sociales et de Santé
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PANJO
Record Dates: First submitted 2016-12-02; First posted 2017-01-02 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Parent-Child Relations; Maltreatment by Parent; Parents; Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PANJO Intervention (Experimental): 201 nulliparous women will be recruited within the PMI public services. Nurses/Midwives will propose to enroll in the PANJO group, which consist in receiving 6 to 12 home visits by a home visitor trained by the PANJO team The visits will consist on 45 to 90-minutes interventions aiming at supporting the family in the everyday challenges they may encounter, and to support the development of qualitative parent-child relationships.
  Interventions: Other: PANJO
- Service as usual (Active Comparator): 246 nulliparous women will be recruited within several maternity wards. They will recieve the services they may request from (a) the maternities, (b) the maternal and child protection services (PMI, usually 1 or 2 home visit without any standards) or any other service available. They will be provided with the address and telephone of the closest maternity ward.
  Interventions: Other: PANJO

INTERVENTIONS:
Other: PANJO — PANJO consists on a 6 to 12 home visitation intervention aiming at supporting the parents, supporting their upcoming then relationship with their first newbord child and to help them reaching all services they may need.

SUMMARY:
The PANJO study aims to evaluate, within the French public health services, the impact of a home visitors training on parent-child attachment, families outcomes, use of services and child maltreatment indicators.

DETAILED DESCRIPTION:
In translation

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Pregnant <32 weeks of amenorrhea
* Answers yes to the following question: "do you feel alone facing the upcoming changes related to your child"

Exclusion Criteria:

* Intends to move outside the area in which she can receive the intervention
* Sees a psychologist or psychiatrist at least once per week
* Refuses to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2016-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Parental self-efficacy | Child 6th month
  20-item questionnaire parental evaluating parental self efficacy and coercitive behaviors
Parental Stress Inventory | Child 6th month
  Subscale "parent-child interactions"
Service Use | Child 6th month
  Use of all social and health services by families
Accidents | Child 6th month
  Nb of accidents and accidents leading to hospitalization in children
Child Maltreatment | Child 6th month
  Number of services required within the child protection services

SECONDARY OUTCOMES:
Pacotis-Parental Impact | Child 6th and 12th month
  Subscale of parental impact self-reported
Parental Stress Inventory - Parental Distress | Child 6th and 12th month
  Measure of Parental Distress
Knowledge of Infant Development Inventory (KIDI questionnaire) | Child 6th and 12th month
  Measure of Knowledge of Infant Development
Edinburgh Postnatal Depression Scale | Child 6th and 12th month
  Measure of depression in mothers

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Saïas, Ph.D., Principal Investigator — L'Agence des Nouvelles Interventions Sociales et de Santé
Locations (1):
- Agence Nationale de Santé Publique, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saïas, T, Delawarde, C, Colson, S, Planche, M, Vallée, V, Du Roscoät, E, Bonnard, A, Bodard, J, Dugravier, R. De l'expérimentation scientifique à l'implantation dans les services publics : le projet Panjo. Revue Francophone Internationale de Recherche Infirmière, 2 : 232-241, 2016.